CLINICAL TRIAL: NCT06040710
Title: Artificial-intelligence-based QUAntification of Size measuremeNts of Adenoma in Routine Endoscopy
Acronym: AQUASNARE
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AI02
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Polyp; Colorectal Adenoma
Keywords: Polyp Size; Colorectal Polyp; Artificial Intelligence; Endoscopy; Follow-up interval

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Intervention arm: All patients within the study are included in the intervention arm: polyp detected within these patients will be measured according to the study protocol using two different methods.
  Interventions: Device: POSEIDON size estimation software with the EndoMind polyp detection system

INTERVENTIONS:
Device: POSEIDON size estimation software with the EndoMind polyp detection system — Polyp size estimation using the POSEIDON software and bounding boxes of the EndoMind polyp detection system.

SUMMARY:
Polyp size and count determines the follow-up intervals after colonoscopy. However, relying on the endoscopist's optical diagnosis for size estimation has shown considerable variability, leading to erroneous surveillance intervals and increased colorectal cancer risk. This study aims to assess the effectiveness of a new polyp size estimation software, called POSEIDON, which uses the tip of the auxiliary water-jet as reference and is implemented together with the EndoMind polyp detection system.

DETAILED DESCRIPTION:
Objective:

The primary aim of this study is to conduct a superiority analysis between POSEIDON and endoscopist optical estimation, focusing on the errors of polyp size measurement. Secondary objectives encompass subgroup analyses concerning varying polyp sizes and histology, potential impact on follow-up protocols based on polyp sizes, and determination of the percentage of cases where obtaining measurements with POSEIDON proves unfeasible.

Study Design:

Single center, endoscopist blinded study. Considering the results of the preliminary study, a total of 42 pairs of measurements suffices to extrapolate statistical significance for a power of 90% and a significance level of 0.05. Taking dropout rates, average number of polyps per patient, polyp detection rate, the number of patients expected to be enrolled for the study is 156. For obtaining the gold standard measurement, images from the examination recording where the tip of a snare is placed next to the polyp are extracted. The snare tip and polyp are manually segmented and their largest diameter in pixels is manually calculated. The diameter of the snare-tip will be measured after the examination to account for production based variations. Based on this, the gold standard polyp size is calculated.

AI setup and limitations:

The version of the polyp detection system, EndoMind, is an updated version of the one published in (PMID: 35543874). Notably, the POSEIDON method has undergone dual refinements from its first published version (PMID: 37080235). Firstly, the AI model for water-jet tip detection has been further trained using images from colonoscopy videos, leading to performance improvements. Secondly, the pixel-to-millimeter conversion methodology has been optimized to align with the specifications of the endoscopes employed in the trial.

To obtain a polyp size estimation, initially the polyp is detected by means of a bounding box through the EndoMind system. Then, once water-jet is sprayed next to the polyp, POSEIDON detects the tip of the water-jet, where it touches the mucosa. The coordinates of the tip in the endoscopic image are correlated to the distance of the endoscope to the mucosa. With the above, the largest diameter of the bounding box is converted from pixels to millimeters, resulting in the size estimation.

For measurement acquisition, the system is initiated at the beginning of the examination and deactivated at its conclusion, facilitated by a dedicated button press. Concerning expert-system interaction, the CADe system's identifications consistently appear on an auxiliary screen within the endoscopist's workspace. On this screen, precise visualization of the impact point between the water-jet beam and the mucosa follows water-jet detection. Subsequently, the endoscopist receives visual affirmation of a successful calculation of polyp size estimation, derived from the bounding box on the screen. The endoscopist evaluates the alignment of this box around the polyp to assess the accuracy measurement outcome. Importantly, throughout these operations, the endoscopist remains blinded to the size estimated by POSEIDON. The endoscopist also reports polyp cases where they are unable to obtain a proper measurement.

Study population:

All adult patients with screening or surveillance colonoscopies that do not match the exclusion criteria will be asked for informed consent.

Intervention:

Upon polyp identification by the endoscopist, the visual assessment will be conducted, followed by obtaining a satisfactory measurement using POSEIDON when possible, as described in the AI methods section. To eliminate potential learning bias and optimize efficiency, the examiner will be blinded to the immediate measurement result. Finally, after both measurements are obtained, an instrument tip of known size will be positioned adjacent to the polyp, which is to be later used for obtaining the gold-standard polyp size.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Scheduled for colonoscopy

Exclusion Criteria:

Patient Level:

* Inflammatory Bowel Disease
* Familiar Polyposis Syndrome

Data Level

* Failure to initialize system before examination
* Missing image instrument placed next to polyp to obtain gold standard

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years), scheduled for screening, surveillance, or diagnostic colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Error of size estimation for colorectal polyps using POSEIDON versus physician optical evaluation | Through study completion, an average of 5 months
  The error between gold standard polyp size and estimation using POSEIDON and optical estimation will be compared in pairs for the same polyps.

SECONDARY OUTCOMES:
Error of size estimation for colorectal polyps using POSEIDON versus physician optical evaluation for different size categories | Through study completion, an average of 5 months
  Polyps will be split into size categories based on national and international guidelines. The study will assess the errors of both POSEIDON and optical estimation within each group through pairwise comparison
Error of size estimation for colorectal polyps using POSEIDON versus physician optical evaluation for polyps with different histologies | Through study completion, an average of 5 months
  Polyps will be split into based on their histological evaluation. The study will assess the errors of both POSEIDON and optical estimation within each group through pairwise comparison.
Rate of change in guideline-suggested follow-up interval based purely on detected polyp size. | Through study completion, an average of 5 months
  The study determines follow-up intervals based on three international standards, solely considering polyp size estimated by the two methods.
Percentage of polyps where endoscopists failed to obtain POSEIDON measurement. | Through study completion, an average of 5 months
  Evaluation of the percentage polyps for which the endoscopist was unable to obtain a proper measurement with the proposed method.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lux TJ, Banck M, Sassmannshausen Z, Troya J, Krenzer A, Fitting D, Sudarevic B, Zoller WG, Puppe F, Meining A, Hann A. Pilot study of a new freely available computer-aided polyp detection system in clinical practice. Int J Colorectal Dis. 2022 Jun;37(6):1349-1354. doi: 10.1007/s00384-022-04178-8. Epub 2022 May 11. PMID 35543874
- [Background] Sudarevic B, Sodmann P, Kafetzis I, Troya J, Lux TJ, Sassmannshausen Z, Herlod K, Schmidt SA, Brand M, Schottker K, Zoller WG, Meining A, Hann A. Artificial intelligence-based polyp size measurement in gastrointestinal endoscopy using the auxiliary waterjet as a reference. Endoscopy. 2023 Sep;55(9):871-876. doi: 10.1055/a-2077-7398. Epub 2023 Apr 20. PMID 37080235